CLINICAL TRIAL: NCT00388700
Title: Open-Label, Phase 2 Study of GM-CT-01 When Added to a Regimen of Leucovorin, 5-FU, and Avastin as First Line Treatment for Locally Advanced, Unresectable or Metastatic Colorectal Cancer in Subjects Unable to Tolerate Intensive Chemotherapy
Brief Title: A New Agent GM-CT-01 in Combination With 5-FU, Avastin and Leucovorin in Subjects With Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Financing and re-organization
Sponsor: Galectin Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAVFU006
Record Dates: First submitted 2006-10-13; First posted 2006-10-17 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer, DAVANAT, colon cancer, 5-FU
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — galactomannan; Fluorouracil; Leucovorin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GM-CT-01 (Experimental)
  Interventions: Drug: GM-CT-01; Drug: 5-Fluorouracil, Leukovorin, bevacizumab

INTERVENTIONS:
Drug: GM-CT-01 — On Day 1 and 2 of each cycle, GM-CT-01 280 mg/m2 administered IV over 30 minutes with 5-FU (400 mg/m2), followed by a 22-hour continuous infusion of GM-CT-01 (280 mg/m2) with 5-FU (600 mg/m2 .)
  Other Names: DAVANAT
Drug: 5-Fluorouracil, Leukovorin, bevacizumab — On Day 1 and 2 of each cycle, LV (200 mg/m2) will be administered IV over 2 hours, followed by 5-FU 400 mg/m2 in solution with GM-CT-01 280 mg/m2 administered over 30 minutes, followed by a 22-hour continuous infusion of GM-CT-01 (280 mg/m2) and 5-FU (600 mg/m2 ). on Day 3 Avastin® (5 mg/kg)will be given IV over 30 to 90 minutes per the package insert.
  Other Names: 5-FU, LV, Avastin®

SUMMARY:
The purpose of this clinical trial is to determine whether the combination of 5-fluorouracil (5-FU) plus a DAVANAT (carbohydrate polymer) along with Avastin and Leucovorin (LV) is beneficial in treating colorectal cancer in patients unable to tolerate intensive chemotherapy.

DETAILED DESCRIPTION:
This is a Phase II, multi-center study of DAVANAT which has been shown to increase the anti-tumor activity of 5-FU in mice. 5-FU is a chemotherapy drug commonly used to treat tumors. A Phase I study of 40 patients showed that DAVANAT in different doses plus 5-FU was well tolerated in patients with different types of solid tumors who failed standard, approved treatments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Histologically confirmed, unresectable, locally advanced or metastatic colorectal adenocarcinoma (stage III and IV), not amenable to curative surgery or radiotherapy.
* Intolerant of oxaliplatin and/or irinotecan, as demonstrated by unacceptable toxicity after a trial of these agents as first-line therapy, or in the opinion of the Investigator, be judged at high risk for unacceptable toxicity to oxaliplatin and/or irinotecan,
* Presence of at least 1 measurable lesion,
* Have a life expectancy of at least 4 months.
* Women of childbearing potential, have a negative serum pregnancy test at screening and Day 1 treatment and agree to practice abstinence or use an effective method of contraception.

Exclusion Criteria:

* Central nervous system metastasis.
* Bony metastasis as the sole metastasis.
* Received any prior first-line chemotherapy for colorectal cancer.
* Previously exposed to DAVANAT® or Avastin®.
* Known or clinically suspected infection with HIV.
* Participated within 30 days or will participate concurrently in another investigational drug or vaccine study.
* History of drug or alcohol dependence in the past 3 years.
* Other serious, non-malignant, significant, acute or chronic medical or psychiatric illness that in the judgment of the Investigator could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Primary Outcomes: Assess the efficacy and safety of GM-CT-01 administered with 5-FU, LV, and Avastin® in the first-line treatment of unresectable, locally advanced, and/or metastatic CRC. | When 17 evaluable patients will complete the study
  To assess the clinical benefit of a regimen of GM-CT-01/5-FU, LV plus Avastin® when administered intravenously as a first-line treatment to patients with Stage III or IV ,advanced or metastatic CRC. Clinical activity will be assessed by determining the percentage of subjects exhibiting an objective response (complete response [CR]) plus partial response [PR]). Tumor response will be assessed following Response Evaluation by RECIST guidelines.

SECONDARY OUTCOMES:
To evaluate the safety of the DAVANAT®/5-FU, LV plus Avastin® regimen. | Throughout the study and when 17 evaluable patients will when complete the study
  Assess safety of regimen and also patient reported outcomes using a Quality of Life (QoL) instrument.
Explore progression-free survival (PFS) and survival | When at least 17 evaluable patients complete the study
  To explore time to tumor progression, duration of response and and survival at 6 and 12 months after the first dose of study drug.

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (4):
  - Rambam Medical Center, Haifa
  - Kaplan MC, Rehovot
  - Sourasky Medical Center, Tel Aviv
  - Sheba MC, Tel Litwinsky